CLINICAL TRIAL: NCT03188328
Title: A Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, Dosimetry, Maximum Tolerated Dose and Preliminary Efficacy of Intra-lesionally Injected AvidinOX, Followed by Systemic IV Administration of Escalating Doses of [177Lu]DOTA-biotin in Patients With Solid Tumors or Lymphomas With Injectable Neoplastic Lesions.
Brief Title: Safety, Tolerability, PK, Dosimetry, MTD and Preliminary Efficacy of Intra-lesionally Injected AvidinOX, Followed by IV Escalating Doses of [177Lu]DOTA-biotin in Pts With Injectable Solid Tumors or Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AvOX/ST2210-CR-15-001
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Inoperable Solid Tumors or Lymphomas
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AvidinOX/177Lu-ST2210 (Experimental): Patients will receive an intralesion injection of AvidinOX followed by two intravenous infusions of 177Lu- ST2210 with a distance of 14 days between them
  Interventions: Drug: AvidinOX; Drug: 177Lu-ST2210

INTERVENTIONS:
Drug: AvidinOX — AvidinOX vial containing 22.5 mg AvidinOX
  + vials containing 10 ml of water for injection (WFI) for the reconstitution in a clear solution with an AvidinOX concentration of 3 mg/ml. One Intralesion administration of a volume of reconstituted AvidinOX equal to about 15 % of the estimated lesion volume
Drug: 177Lu-ST2210 — 177Lu-ST2210 dose starting at 7.5 Gigabequerel (GBq) ±10%with escalation steps of 2.5 GBq up to 15 GBq ±10%, approximately 1 mg ST2210
Drug: 177Lu-ST2210 — Second dose of 177Lu-ST2210 dose (14 days after the first dose) starting at 7.5 Gigabequerel (GBq) ±10%with escalation steps of 2.5 GBq up to 15 GBq ±10%, approximately 1 mg ST2210

SUMMARY:
Local treatment of unresectable tumors is challenging, particularly with radioactivity. Current practice relies on external beam irradiation or on a variety of medical devices for brachytherapy. Both approaches proved useful in controlling tumor growth but are characterized by poor patient's compliance, significant side effects, high costs and technological complexity hampering wide-spread use. The use of AvidinOX for radionuclide therapy of inoperable cancer lesions will offer a number of advantages compared to current brachytherapy. In fact, the perfusion of a target tissue with AvidinOX, compared to current devices, will allow adapting the therapy to the tumor/organ shape, and it will also make it possible to delay the administration of radioactivity for several days which, according to pre-clinical studies, might be also divided up into repeated doses. AvidinOX linking stably to tissue proteins, does not exhibit the problem of seed migration which is associated with high morbidity. Based on previous findings with AvidinOX in combination with radionuclides in pre-clinical studies as well as data from the clinical use in liver metastases, it can be assumed that intralesional injections of AvidinOX followed by intravenous injections of 177Lu-ST2210 could be a safe and efficacious method for treating inoperable tumor lesions.

DETAILED DESCRIPTION:
The primary objectives of this study are:

1. To identify the Maximum Tolerated Dose (MTD) of two consecutive repeated IV 177Lu-ST2210 administration following a previous tumor intra-lesion/s injection of AvidinOX.
2. To assess safety and tolerability of intra-lesionally injected AvidinOX + IV injected 177Lu-ST2210
3. To evaluate intra-lesional distribution and retention of {AvidinOX + 177Lu-ST2210}-complex in tumor lesion/s
4. To evaluate systemic biodistribution and pharmacokinetics of 177Lu-ST2210 and {AvidinOX + 177Lu-ST2210}- complex

Main secondary objectives are:

1. To evaluate whole body dosimetry of IV 177Lu-ST2210 after prior AvidinOX injection (radiation safety dosimetry)
2. To record individual tumor dosimetry
3. To evaluate preliminary efficacy of {AvidinOX + 177Lu-ST2210}-complex in reducing tumor size and metabolic activity.
4. To evaluate damage of tumor cells by radioactivity and immunogenic cell death
5. To evaluate whole body safety dosimetry and dose linearity
6. To evaluate pharmacokinetics of ST2210 in plasma and urine

ELIGIBILITY:
Main Inclusion Criteria:

* Presence of inoperable tumor lesion/s from histologically confirmed solid tumors or lymphomas, in patients with at least one lesion ≥ 1 cm and suitable for intra-lesional injection, who have disease progression after treatment with available therapies, or who are intolerant to such treatments
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* If the patient received previous radiation therapy, the total absorbed radiation dose at the bone marrow level must be ≤ 1 Gy
* Life expectancy of at least 3 months
* Total tumor burden requiring ≤ 75 mL AvidinOX injection
* Clotting parameters within normal limits or maximum 25% outside of the the normal ranges
* Haematological and liver function test results ≤ grade 2 toxicity (according to US National Cancer Institute's Common Terminology) Criteria for Adverse Events v4.03 [CTCAE
* Urine protein (dipstick): negative or trace; in case of trace, a urinalysis has to be performed in the local laboratory and have to confirm that such abnormality is not to be considered clinically significant, according to the investigator's judgement
* Creatinine ≤ 1.7 mg/dL
* eGFR> 60% of mean age adjusted normal values
* Written informed consent

Main Exclusion Criteria:

* Known hypersensitivity to Avidin or AvidinOX (e.g. hen egg)
* Known hypersensitivity to ST2210 (DOTA biotin) or any excipient.
* Presence of unreachable (e.g. located in a region that cannot be reached by needle) or untreatable tumor lesions so that the benefit from the treatment of the treatable lesions does not justify patient's inclusion
* Active infection at screening or history of severe infection within the previous 3 months, if clinically relevant at screening as considered by the investigator
* Known human immunodeficiency virus (HIV) positive serology or chronically active hepatitis B or C.
* Administration of another investigational medicinal product within 30 days before the screening period.
* Patient who underwent chemotherapy, radiation therapy within 15 days before the screening period
* Previous treatment with any radiopharmaceutical within a period corresponding to 8 half-lives of the radionuclide used for labeling the respective radiopharmaceutical prior to the administration of study drug.
* Women of child-bearing potential without a serum negative pregnancy test and not willing to refrain from sexual activity or to utilize an adeguate contraceptive methods during all the course of the study
* Men unwilling to use appropriate contraceptive methods during the study and up to six months follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity evaluated using NCI Common Toxicity Criteria (CTCAE 4.03) | Up to six weeks after the second 177Lu-ST2210 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Subbiah, MD, Principal Investigator — Dep. of Investigational Cancer Therapeutics - U. T. M. D. Anderson Cancer Center
Locations (1):
- Dep. of Investigational Cancer Therapeutics - U. T. M. D. Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vesci L, Carollo V, Rosi A, De Santis R. Therapeutic efficacy of intra-tumor AvidinOX and low systemic dose biotinylated cetuximab, with and without cisplatin, in an orthotopic model of head and neck cancer. Oncol Lett. 2019 Mar;17(3):3529-3536. doi: 10.3892/ol.2019.10003. Epub 2019 Feb 1. PMID 30867794